CLINICAL TRIAL: NCT04247529
Title: Effects of Prior Exposure to Conflicting Health Information on Responses to Subsequent Unrelated Health Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019NTLS140; R21CA218054 (NIH)
Record Dates: First submitted 2020-01-16; First posted 2020-01-30 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Communication Research

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No exposure to conflict (Placebo Comparator)
  Interventions: Other: No exposure to conflicting health information
- Exposure to conflict (Experimental)
  Interventions: Other: Exposure to conflicting health information

INTERVENTIONS:
Other: Exposure to conflicting health information — At 2 time points across a ~28-day period, participants will be exposed to news stories and social media posts about 6 health topics: mammography screening, prostate-specific antigen (PSA) testing, Vitamin D supplementation, carbohydrate consumption, alcohol consumption, and breastfeeding. Participants in the conflict (experimental) group will have conflicting information added to these news and social media posts.
  Arms: Exposure to conflict
Other: No exposure to conflicting health information — At 2 time points across a ~28-day period, participants will be exposed to news stories and social media posts about 6 health topics: mammography screening, prostate-specific antigen (PSA) testing, Vitamin D supplementation, carbohydrate consumption, alcohol consumption, and breastfeeding. Participants in the no conflict (comparator) group will have no conflicting information included in these news and social media posts.
  Arms: No exposure to conflict

SUMMARY:
Many population-level public health strategies-including media campaigns and other behavioral interventions, screening recommendations, and vaccination policies-rely on messaging to promote cancer prevention and control. These strategies do not take place in a vacuum; rather, they occur in the context of a broader public information environment, which is increasingly characterized by conflicting and often controversial health information. Although studies have documented that such information is prevalent, a critical question remains unanswered: does exposure to conflicting health information in people's routine interactions with the broader information environment threaten the success of message-based population-level public health strategies? And, if so, who is most susceptible to the effects of such exposure? This study will provide a rigorous empirical test of these critical answered questions, guided by two specific aims: First, to evaluate whether prior exposure to conflicting health information influences responses to subsequent unrelated and uncontested health messages, a phenomenon that has been described as "carryover effects" (Primary Aim); and second, to identify whether there are individual-level differences in how conflict affects responses to these unrelated and uncontested health messages (Secondary Aim).

DETAILED DESCRIPTION:
To accomplish these aims, an online survey-based experiment using a population-based sample of U.S. adults (anticipated N=1,800) will be conducted. At 2 time points across a 28-day period, participants will be exposed to news stories and social media posts about 6 health topics: mammography screening, prostate-specific antigen (PSA) testing, Vitamin D supplementation, carbohydrate consumption, alcohol consumption, and breastfeeding. Participants will be randomized to 1 of 2 treatment groups that differ only in the amount of conflict presented in these news and social media posts (conflict, no conflict). At a third time point, after the exposure to conflict period, all participants will be exposed to 3 (out of a possible 9) messages from existing health campaigns about 3 behaviors for which there is scientific consensus: fruit and vegetable consumption, colorectal cancer screening, and physical activity. To assess carryover effects (Primary Aim), participants' receptivity to these messages-as measured through several affective and cognitive responses (e.g., confidence in the evidence presented)-will be measured. Message receptivity is expected to be lower among those who were randomized to receive conflicting health information. Individual-level differences in message receptivity are possible; thus exploratory analyses (Secondary Aim) will be conducted to assess whether carryover effects of exposure to conflict may be more pronounced among certain groups (e.g., those with greater trust in media sources, those of lower socioeconomic position).

ELIGIBILITY:
Inclusion Criteria:

* 18+ U.S. adults
* Members of NORC's AmeriSpeak Panel (https://amerispeak.norc.org/Pages/default.aspx)
* Able to complete web-based survey
* Able to read in English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6046 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Negative affective responses | Up to 42 days
  * Participants are asked to indicate how "the ad you just saw made you feel"
  * 7 affective responses are randomly ordered: interested, frustrated, surprised, annoyed, distressed, optimistic, worried (response options: 1 "very slightly or not at all" to 5 "extremely")
Counterarguing | Up to 42 days
  • Participants are asked to indicate the extent to which they agree or disagree with 4 statements (randomly ordered; response options: 1 "strongly disagree" to 5 "strongly agree"):
  * "I found myself agreeing with the ad" (reverse coded)
  * "I thought of points that went against what the ad was saying"
  * "I accepted the ad's claims" (reverse coded)
  * "While reading the ad, I was skeptical of its claims"
Reactance/threat to freedom | Up to 42 days
  • Participants are asked to indicate the extent to which they agree or disagree with the following statement (response options: 1 "strongly disagree" to 5 "strongly agree"): "I felt like the ad was trying to manipulate me"
Other negative cognitive responses to ad claims | Up to 42 days
  • Participants are asked to indicate whether "the claims in the ad I just saw are" (randomly ordered; response options: 1 "strongly disagree" to 5 "strongly agree"): exaggerated, flawed, believable (reverse coded), reasonable (reverse coded)
Perceived argument strength | Up to 42 days
  • Participants are asked to indicate the extent to which they agree or disagree with 2 statements (randomly ordered; response options: 1 "strongly disagree" to 5 "strongly agree"):
  * "The ad was convincing"
  * "The ad gave me a strong reason to [engage in the behavior specified in the ad]"
Response efficacy | Up to 42 days
  • Participants are asked to respond to two items, presented in random order:
  * "How confident are you that there is evidence to support the ad's claims?" (1 "not confident at all" to 7 "extremely confident")
  * "How much do you think your health would benefit if you [engaged in the behavior specified in the ad]?" (1 "not at all" to 7 "extremely")

CONTACTS AND LOCATIONS:
Locations (1):
- NORC at the University of Chicago (online only), Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Within one year of study completion, the final, cleaned, de-identified study dataset may be made available to third-party users under a data-sharing agreement that provides for: 1) a commitment to using the data only for research purposes; 2) a commitment to securing the data using appropriate information technology; and 3) a commitment to destroying or returning the data after analyses are completed. Requests for data sharing will be considered by the investigator team via in-person meetings and approved by consensus; meeting minutes will be taken to ensure transparent decision making and conflict of interest avoidance.